CLINICAL TRIAL: NCT07347730
Title: Clinical Study of Myofascial Trigger Points(MTrPs) Injection in the Treatment of Chronic Musculoskeletal Pain(CMP), Chronic Migraine and Cervicogenic Headache
Brief Title: Clinical Study of Myofascial Trigger Points(MTrPs) Injection in the Treatment of Chronic Cervicogenic Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director, Department of Pain Management, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2025-317-02-05
Record Dates: First submitted 2025-12-28; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Myofascial Trigger Points; Cervicogenic Headache; Dorsal Root Ganglion
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTrPs injection group (Experimental): MTrPs injection with triamcinolone acetonide.
  Interventions: Procedure: MTrPs injection
- C2 dorsal rami block group (Active Comparator): C2 dorsal rami block with triamcinolone acetonide.
  Interventions: Procedure: C2 dorsal root ganglion blocks

INTERVENTIONS:
Procedure: MTrPs injection — The volume of infiltration solution is determined by the number of trigger points, with each trigger point receiving 1 mL of injection volume. The injection solution is prepared by combining 1 mL of triamcinolone acetonide (40 mg/mL), lidocaine, and normal saline, resulting in a final lidocaine concentration of 1%. A 25-gauge needle is used to inject perpendicular to the skin surface at the selected tender points, with the solution administered as a single bolus into each tender point within 10 seconds.
  Arms: MTrPs injection group
Procedure: C2 dorsal root ganglion blocks — Patients in the nerve block group received ultrasound-guided bilateral dorsal root ganglion blocks of C2 spinal nerve. The injection solution was prepared using 1 ml of 2% lidocaine and 1 ml of triamcinolone acetonide (40 mg/mL), with a volume of 1 ml administered per side.
  Arms: C2 dorsal rami block group

SUMMARY:
Chronic cervicogenic headache is a common disease in China, with a high incidence among the elderly, and has a significant impact on patients' quality of life. Currently, both domestic and international studies have confirmed that glucocorticoid injection at myofascial trigger points(MTrPs) can alleviate patients' pain symptoms. MTrPs injection is safe and easy to operate, and can improve the clinical management efficiency of patients with chronic cervicogenic headache. Therefore, we designed a prospective, randomized controlled, blinded outcome, non-inferiority study to compare the long-term clinical efficacy of glucocorticoid injection at myofascial trigger points and greater occipital nerve block injection in treating chronic cervicogenic headache. Patients will be randomly divided into two groups and receive either glucocorticoid injection at MTrPs or dorsal rami blocks of C2 spinal nerves. After treatment, patients will be followed up for 2 years. Their NRS scores, attack frequency, attack duration, HIT-6 scores, Patient Global Impression of Change(PGIC) scale, and adverse reactions will be recorded at 2 weeks, 4 weeks, 8 weeks, 12 weeks, and 24 weeks. If the results indicate that the clinical efficacy of myofascial trigger point injection for chronic cervicogenic headache is not inferior to that of injection at intra-articular injection, it will provide a safe and simple treatment option that is easy to promote for patients who do not respond to conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervicogenic headache by at least two pain specialists or neurologists;
* Disease duration of at least 3 months;
* Age between 18 and 65 years;
* Numerical Rating Scale (NRS) score ≥ 3 despite conservative pharmacological treatment;
* Signed informed consent form.

Exclusion Criteria:

* History of allergy to trial medications such as corticosteroids;
* Alcohol abuse; long-term use of opioids (exceeding 2 weeks or more than 3 days per week for over 1 month); suspected use of sedative or analgesic medications; patients on long-term steroid therapy;
* Severe neurological disorders, significant hepatic or renal dysfunction, heart failure, coagulation abnormalities, gastric ulcer, diabetes, inflammatory rheumatic diseases, etc.;
* Inability to use pain assessment scales;
* Presence of local or systemic infection;
* Pregnant or lactating patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
NRS pain scores | at the 4-weeks
  The pain intensity of the headache will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.

SECONDARY OUTCOMES:
NRS pain scores | at the 2, 4, 8, 12, and 24 weeks
  The pain intensity of the headache will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
Attack frequency and duration | at the 2, 4, 8, 12, and 24 weeks
  The frequency of headache and its duration
The Patient Global Impression of Change (PGIC) scale | at the 2, 4, 8, 12, and 24 weeks
  The Patient Global Impression of Change (PGIC) scale is a patient-rated instrument used to evaluate overall change in status following treatment. It employs a 7-point Likert scale (1 = "very much worse" to 7 = "very much improved"), focusing on the patient's subjective perception of symptoms, function, and quality of life. The evaluation criterion defines a score of 5 or higher as indicative of "improvement" (mild/moderate/marked), a score of 4 as "no change," and scores of 3 or below as "worsening."
Adverse Reactions | Through study completion, an average of 1 year
  Any systemic adverse reactions related to corticosteroids such as hyperglycemic reactions, infection and bleeding at the puncture site.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes